CLINICAL TRIAL: NCT02248974
Title: Development and User Testing of a Decision Aid for Left Ventricular Assist Device (LVAD) Placement
Brief Title: Development & Testing of a Decision Aid for LVAD Placement
Acronym: VADDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other); INTEGRIS Baptist Medical Center (Other); Texas Heart Institute (Other); Wake Forest University Health Sciences (Other); The Cleveland Clinic (Other); Patient-Centered Outcomes Research Institute (Other); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Jennifer Blumenthal-Barby, Assistant Professor of Philosophy/Bioethics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-34286; CDR-1306-01769 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: End-Stage Heart Failure; Bridge-to-Transplant LVAD Placement (BTT); Destination Therapy LVAD Placement (DT); Refusal of LVAD Placement (Decliners); LVAD Caregivers
Keywords: End-Stage Heart Failure; Left Ventricular Assist Device; Decision Aid; Medical Decision-Making

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LVAD Decision Aid (Active Comparator): Decision aid presented to subjects was developed from patient and clinician feedback to increase patient knowledge on the risks, benefits, misconceptions or mispredictions regarding LVADs to help patients make an informed decision on accepting or declining LVAD placement.
  Interventions: Other: LVAD Decision Aid
- No LVAD Decision Aid (No Intervention): The standard education processis institution-specific and unstandardized. The education consists of viewing education pamphlets that are created by device manufacturers. The traditional informed consent process may also include viewing and manipulating the actual device and meeting a patient with a device already implanted. Additionally, the LVAD coordinator describes the device and answers any questions LVAD candidates have.

INTERVENTIONS:
Other: LVAD Decision Aid — Decision aids are interventions or tools designed to facilitate shared decision making and patient participation in health care decisions.
  This Decision Aid was designed to discuss treatment options for patients in end-stage heart failure (i.e LVAD PLACEMENT, PALLIATIVE and SUPPORTIVE CARE).
  Arms: LVAD Decision Aid

SUMMARY:
The goal of this project is to develop a patient-centered decision aid for decision-making about end-stage heart failure treatment. This study seeks to create a decision aid that presents outcomes, risks, projected experiences, and uncertainties about Left Ventricular Assist Device (LVAD) placement to help patients make values-based decisions about placement. The investigators propose a mixed methods design involving a literature search of clinical evidence, semi-structured patient interviews, and quantitative data from a multi-site trial of patients receiving the decision aid compared to patients not receiving the aid.

ELIGIBILITY:
Inclusion Criteria:

* LVAD Candidates (NYHA Class III and IV patients with an acceptable surgical risk/benefit ratio for LVAD implantation and with good psychosocial support, coping mechanisms, and financial resources, as determined by "clearance" from the transplant social worker)
* LVAD Patients
* LVAD Decliners
* LVAD Caregivers

Exclusion Criteria:

* subjects who lack the capacity to give informed consent

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Blumenthal-Barby, PhD, Principal Investigator — Baylor College of Medicine; Kristin M Kostick, PhD, Study Director — Baylor College of Medicine
Locations (7):
- United States (7):
  - Ochsner Health System, New Orleans, Louisiana
  - Cleveland Clinic, Cleveland, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - CHI ST. Luke's - Baylor St. Lukes Medical Center / Texas Heart Institute, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Background] Bruce CR, Delgado E, Kostick K, Grogan S, Ashrith G, Trachtenberg B, Estep JD, Bhimaraj A, Pham L, Blumenthal-Barby JS. Ventricular assist devices: a review of psychosocial risk factors and their impact on outcomes. J Card Fail. 2014 Dec;20(12):996-1003. doi: 10.1016/j.cardfail.2014.09.006. Epub 2014 Sep 17. PMID 25239054
- [Background] Blumenthal-Barby, J. S., Kristin M. Kostick, Estevan D. Delgado, Robert J. Volk, Holland M. Kaplan, L. A. Wilhelms, Sheryl A. McCurdy, Jerry D. Estep, Matthias Loebe, and Courtenay R. Bruce.
- [Derived] Kostick KM, Bruce CR, Minard CG, Volk RJ, Civitello A, Krim SR, Horstmanshof D, Thohan V, Loebe M, Hanna M, Bruckner BA, Blumenthal Barby JS, Estep JD. A Multisite Randomized Controlled Trial of a Patient-Centered Ventricular Assist Device Decision Aid (VADDA Trial). J Card Fail. 2018 Oct;24(10):661-671. doi: 10.1016/j.cardfail.2018.08.008. Epub 2018 Sep 7. PMID 30195826
- [Derived] Bruce CR, Minard CG, Wilhelms LA, Abraham M, Amione-Guerra J, Pham L, Grogan SD, Trachtenberg B, Smith ML, Bruckner BA, Estep JD, Kostick KM. Caregivers of Patients With Left Ventricular Assist Devices: Possible Impacts on Patients' Mortality and Interagency Registry for Mechanically Assisted Circulatory Support-Defined Morbidity Events. Circ Cardiovasc Qual Outcomes. 2017 Jan;10(1):e002879. doi: 10.1161/CIRCOUTCOMES.116.002879. PMID 28073849
- [Derived] Kostick KM, Minard CG, Wilhelms LA, Delgado E, Abraham M, Bruce CR, Estep JD, Loebe M, Volk RJ, Blumenthal-Barby JS. Development and validation of a patient-centered knowledge scale for left ventricular assist device placement. J Heart Lung Transplant. 2016 Jun;35(6):768-76. doi: 10.1016/j.healun.2016.01.015. Epub 2016 Jan 21. PMID 26922278
- [Derived] Bruce CR, Blumenthal-Barby JS, Meyers D. Benefits and Challenges of Early Introduction of Left Ventricular Assist Device Placement: A Patient-Centered Perspective. J Am Coll Cardiol. 2015 Oct 20;66(16):1762-1765. doi: 10.1016/j.jacc.2015.08.852. No abstract available. PMID 26483098
- [Derived] Blumenthal-Barby JS, Kostick KM, Delgado ED, Volk RJ, Kaplan HM, Wilhelms LA, McCurdy SA, Estep JD, Loebe M, Bruce CR. Assessment of patients' and caregivers' informational and decisional needs for left ventricular assist device placement: Implications for informed consent and shared decision-making. J Heart Lung Transplant. 2015 Sep;34(9):1182-9. doi: 10.1016/j.healun.2015.03.026. Epub 2015 Mar 31. PMID 26087668
- See also: Project Website — http://www.lvaddecisionaid.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled a total of 98 participants. This number is consistent between the Protocol Section and the Participant Flow Module.
Groups:
- LVAD Decision Aid: Decision aid presented to subjects was developed from patient and clinician feedback to increase patient knowledge on the risks, benefits, misconceptions or mispredictions regarding LVADs to help patients make an informed decision on accepting or declining LVAD placement.
  LVAD Decision Aid: Decision aids are interventions or tools designed to facilitate shared decision making and patient participation in health care decisions.
  This Decision Aid was designed to discuss treatment options for patients in end-stage heart failure (i.e LVAD PLACEMENT, PALLIATIVE and SUPPORTIVE CARE).
Period: Baseline
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Started | 47 | 51
Completed | 47 | 51
Not Completed | 0 | 0
Period: 1-Day Follow-Up
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Started | 47 | 0 ("No DA" group did not receive 1-Day Follow-up survey.)
Completed | 37 | 0 ("No DA" group did not receive 1-Day Follow-up survey.)
Not Completed | 10 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Enrolled in another study | 1 | 0
Period: 1-Week Follow-Up
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Started | 37 | 51
Completed | 29 | 34
Not Completed | 8 | 17
Not completed — Became ineligible for LVAD | 4 | 1
Not completed — Enrolled in another study | 1 | 1
Not completed — Transferred to another facility | 1 | 0
Not completed — Cognitive Difficulty | 1 | 0
Not completed — Death | 1 | 1
Not completed — Excluded because of age | 0 | 1
Not completed — Noncompliant with terms of participation | 0 | 1
Not completed — Timing: implanted before survey | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 8
Period: 1-Month Follow-Up
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Started | 29 | 34
Completed | 27 | 31
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid | Total
Number analyzed (Participants) | 47 | 51 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.61 (14.03) | 59.94 (9.67) | 59.77 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 41 | 54
  Male | 34 | 10 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 38 | 43 | 81
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 11 | 27
  White | 29 | 37 | 66
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Caregiver [Count of Participants; unit: Participants]
  0 Caregivers | 0 | 1 | 1
  1 Caregiver | 8 | 16 | 24
  2 Caregivers | 16 | 16 | 32
  >=3 Caregivers | 23 | 16 | 39
  Prefer not to answer | 0 | 2 | 2
Income [Count of Participants; unit: Participants]
  <$15,000 | 14 | 13 | 27
  $15,000-$30,000 | 8 | 10 | 18
  $30,000-$60,000 | 5 | 6 | 11
  $60,000-$100,00 | 5 | 6 | 11
  >$100,000 | 5 | 2 | 7
  Prefer not to answer | 10 | 14 | 24
Marital Status [Count of Participants; unit: Participants]
  Married | 31 | 30 | 61
  Divorced | 5 | 4 | 9
  Separated | 0 | 2 | 2
  Widowed | 4 | 3 | 7
  Single/never married | 7 | 9 | 16
  Common law | 0 | 2 | 2
  Other | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  8th grade or less | 5 | 2 | 7
  Some high school | 8 | 4 | 12
  High school degree/GED | 16 | 18 | 34
  Some college | 8 | 16 | 24
  4-yr college graduate | 4 | 7 | 11
  Prefer not to answer | 6 | 3 | 9
  Missing data | 0 | 1 | 1
Insurance [Count of Participants; unit: Participants]
  Private | 16 | 22 | 38
  Public | 15 | 14 | 29
  Private and Public | 14 | 10 | 24
  Prefer not to answer | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Assist Device (LVAD) Knowledge Scale
Description: Questionnaire measuring subject's knowledge about Left Ventricular Assist Device therapy. Knowledge is reported on a scale from 1-100, with higher scores indicating greater knowledge. At Baseline, this scale measures LVAD knowledge before patients receive any formal education (from their LVAD coordinators and/or physicians) about LVAD therapy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No LVAD Decision Aid: The standard education process is institution-specific and unstandardized. The education consists of viewing education pamphlets that are created by device manufacturers. The traditional informed consent process may also include viewing and manipulating the actual device and meeting a patient with a device already implanted. Additionally, the LVAD coordinator describes the device and answers any questions LVAD candidates have.
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 47 | 51
units on a scale | 45.6 (22.2) | 43.8 (18.3)

2. Primary Outcome: Left Ventricular Assist Device (LVAD) Knowledge Scale
Description: Questionnaire measuring subject's knowledge about Left Ventricular Assist Device therapy. Knowledge is reported on a scale from 1-100, with higher scores indicating greater knowledge. At this time-point, the scale measures LVAD knowledge at 1 week following both formal education (from the clinic) as well as from our decision aid about LVAD therapy.
Time Frame: 1-Week Follow-up
Population: Analysis only includes individuals who responded to the measure at 1-Week Follow-Up (DA=29, no-DA=34, Total=63).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 29 | 34
units on a scale | 67.8 (15.6) | 59.3 (12.4)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; The model uses a general linear mixed model with fixed effects for baseline Knowledge Scale score, time (discrete), arm, and a time-arm interaction term. The matrix of correlated residual terms assumes an unstructured format; Test type: Superiority; p = 0.01, Mixed Models Analysis

3. Primary Outcome: Left Ventricular Assist Device (LVAD) Knowledge Scale
Description: Questionnaire measuring subject's knowledge about Left Ventricular Assist Device therapy. Knowledge is reported on a scale from 1-100, with higher scores indicating greater knowledge. At this time-point, the scale measures LVAD knowledge at 1 month following both formal education (from the clinic) as well as from our decision aid about LVAD therapy.
Time Frame: 1-Month Follow-up
Population: Analysis only includes individuals who responded to the measure at 1-Week Follow-Up (DA=27, no-DA=31, Total=58).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 31
units on a scale | 27.9 (5.7) | 22.9 (6.6)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; The model uses a general linear mixed model with fixed effects for baseline KS score, time (discrete), arm, and a time-arm interaction term. The matrix of correlated residual terms assumes an unstructured format; Test type: Superiority; p = 0.47, Mixed Models Analysis

4. Secondary Outcome: Decisional Conflict Scale
Description: Measures the construct of decisional conflict, using a 5-point Likert scale with 12 question items. All question items have a positive valence, with higher scores indicating lower decision conflict. Scores range from 0-100.
Time Frame: Baseline
Population: Analysis includes only those participants who completed the measure at Baseline (DA=44, no-DA=50, Total=94).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 44 | 50
units on a scale | 23.1 (20.7) | 29.3 (19.3)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Used Wilcoxon 2-sample test to see if DA group had significantly better (i.e. lower) Decisional Conflict Scores than no-DA (Control) group; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Decisional Conflict Scale
Description: Measures the construct of decisional conflict (at this timepoint, 1 week after baseline), using a 5-point Likert scale with 12 question items. All question items have a positive valence, with higher scores indicating lower decision conflict. Scores range from 0-100.
Time Frame: 1 Week Follow-up
Population: Analysis includes only those participants who completed the measure at Baseline (DA=29, no-DA=33, Total=62).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 29 | 33
units on a scale | 15.7 (11.8) | 17.4 (14.7)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: collaboRATE-Shared Decision Making
Description: Measures a participant's perceived degree of shared decision-making about treatment (at this time point: 1 week after baseline). All question items have a positive valence (higher scores indicating greater shared decision-making, a more positive outcome), with scores ranging from 0-100.
Time Frame: 1 Week Follow-up
Population: Analysis only includes participants who responded to the measure at 1-Week Follow-Up (DA=28, no-DA=34, Total=62).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 28 | 34
units on a scale | 88.4 (19.3) | 89.6 (15.6)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: collaboRATE-Shared Decision Making
Description: Measures a participant's perceived degree of shared decision-making about treatment (at this time point: 1 month after baseline). All question items have a positive valence (higher scores indicating greater shared decision-making, a more positive outcome), with scores ranging from 0-100.
Time Frame: 1 Month Follow-up
Population: Analysis only includes participants who responded to measure at 1-Month Follow-Up (DA=26, no-DA=31, Total=57).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 31
units on a scale | 90.4 (14.3) | 89.8 (17.2)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Satisfaction With Decision Making Process
Description: Measures a participant's satisfaction with their decision of treatment (at this time point: 1 month after baseline). All question items have a positive valence (higher scores indicating greater satisfaction with the decision making process, a more positive outcome), with scores ranging from 0-100.
Time Frame: 1 Month Follow-up
Population: Analysis only includes participants who responded to measure at 1-Month Follow-Up (DA=26, no-DA=31, Total=67).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 31
units on a scale | 75.6 (23.7) | 76.8 (20.0)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Ottawa Decision Regret Scale
Description: The 'Decision Regret Scale' measures "distress or remorse after a (health care) decision." In a short introductory statement, respondents should be asked to reflect on a specific past decision, and then asked to indicate the extent to which they agree or disagree with the statements in the regret scale by indicating a number from 1 (Strongly Agree) to 5 (Strongly Disagree) that best indicates their level of agreement. Regret is measured at a point in time when the respondent can reflect on the effects of the decision. Items 2 and 4 should be reverse coded so that, for each item, a higher number will indicate more regret. To help others interpret the score more readily with other scales ranging from 0 to 100, these scores can then be converted to a 0-100 scale by subtracting 1 from each item then multiply by 25. To obtain a final score, the items are summed and averaged. A score of 0 means no regret; a score of 100 means high regret.
Time Frame: 1 Month Follow-up
Population: Analysis only includes participants who responded to measure at 1-Month Follow-Up (DA=26, no-DA=31, Total=67).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 31
units on a scale | 11.5 (13.3) | 12.9 (16.6)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Satisfaction With Life Scale
Description: Measures participants' perceived Satisfaction with Life. Out of 0-30 scale. Higher scores indicate higher satisfaction with life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 47 | 51
units on a scale | 22.8 (6.6) | 20.4 (7.2)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Satisfaction With Life Scale
Description: as for outcome 10
Time Frame: 1 Month Follow-up
Population: Analysis only includes participants who responded to measure at 1-Month Follow-Up (DA=26, no-DA=31, Total=67).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 31
units on a scale | 27.9 (6.7) | 22.9 (6.6)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Preparedness for Decision-Making Scale
Description: The Preparedness for Decision-Making Scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation visit and making a health decision (treatment/diagnostic/screening, etc.). Items can be summed and scored (sum the 10 items and divide by 10). B) Scores are converted to a 0-100 scale by: subtracting 1 from the summed score in part a) and multiplying by 25. Higher scores indicate higher perceived level of preparation for decision-making.
Time Frame: 1 Week Follow-up
Population: Analysis only includes participants who responded to measure at 1-Week Follow-Up (DA=27, no-DA=33, Total=60).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 33
units on a scale | 86.9 (15.1) | 81.8 (17.4)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Usability and Acceptability: Helped me Understand More About the Risks and Benefits of Treatment.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: Analysis included only those participants who completed this question in the 1-Day Follow-up measure, which was 35 patients in the DA group. The no-DA group did not receive the measure.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 35 | 0
Participants
  Strongly Agree | 21 | 0
  Agree | 12 | 0
  Neutral | 2 | 0
  Disagree | 0 | 0
  Strongly Disagree | 0 | 0

14. Secondary Outcome: Shared Decision-Making (SDM-9)
Description: A brief patient-report instrument for measuring Shared Decision Making (SDM) in clinical encounters. All question items have a positive valence. Summing up all items leads to a raw total score between 0 and 45. Multiplication of the raw score by 20/9 provides a score forced (transformed) to range from 0 to 100, where 0 indicates the lowest possible level of SDM and 100 indicates the highest extent of SDM. As it is more intuitively interpretable, the authors of the scale encourage the use of the transformed score, which we used.
Time Frame: 1-Week Follow-Up
Population: Analysis only includes participants who responded to measure at 1-Week Follow-Up (DA=27, no-DA=34, Total=61).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 34
units on a scale | 84.8 (16.8) | 84.3 (13.6)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Shared Decision-Making (SDM-9)
Description: as for outcome 14
Time Frame: 1-Month Follow-Up
Population: Analysis only includes participants who responded to measure at 1-Month Follow-Up (DA=25, no-DA=31, Total=56).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 25 | 31
units on a scale | 87.5 (12.8) | 85.2 (15.0)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Number and Percentage of Participants Whose Control Preferences for Treatment Decision-Making Match From Baseline to 1-month Follow-up
Description: Measure of the degree (percentage) of match in patient-reported preferences related to control over treatment decision at Baseline and 1-Month. This data is based on responses to a 1-item questionnaire (i.e. not a scale). Scores are calculated by counting the frequency of matches in patient-reported preferences at two time points. The results are reported as the number of participants with a 1:1 "match" in preferences at both time points.
Time Frame: 1-Month Follow-Up
Population: Analysis only included participants who completed the measure at both Baseline and 1-Month followup, in order to calculate "match" in preferences.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 29 | 25
Participants | 14 | 13

17. Secondary Outcome: Ability to Envision Life With an LVAD: Somewhat/Easy Picturing What to Expect
Description: Percentage of patients reporting that their ability to envision life with an LVAD was "Somewhat Easy" or "Easy."
Time Frame: 1-Week Follow-Up
Population: Analysis only includes those who responded to this measure (DA=27, no-DA =33, Total=60).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 33
Participants | 25 | 25

18. Secondary Outcome: Number and Percentage of Participants Reporting Ability to Envision Life With an LVAD: Difficult/no Idea What to Expect
Description: Number and percentage of patients reporting that their ability to envision life with an LVAD was "Difficult" or that they had "No idea."
Time Frame: 1-Month Follow-Up
Population: Analysis only includes those who responded to this measure (DA=20, no-DA =21, Total=41).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 20 | 21
Participants | 15 | 9

19. Secondary Outcome: Number & Percentage of Participants Who Perceived a Strong Likelihood of Transplant
Description: Measures the number and percentage of participants who perceived a strong likelihood of transplant.
Time Frame: 1-Week Follow-Up
Population: Analysis included only those participants who responded to the measure at 1-week (DA=26, no=DA=33, Total=59).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 33
Participants | 16 | 22
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Number and Percentage of Participants Who Perceived and Strong Likelihood of Transplant
Description: Number and Percentage of participants who perceived and strong Likelihood of Transplant after 1-Month follow-up.
Time Frame: 1-Month Follow-Up
Population: Analysis included only those participants who responded to the measure at 1-month (DA=27, no-DA=31, Total=58).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 31
Participants | 17 | 15
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Participants' Perceived Survival Estimate in Number of Years After LVAD Implant
Description: Patient-reported estimate of number of years the average patient is able to live after LVAD implant. Participants wrote in a number in a blank space, and numbers were recorded.
Time Frame: 1-Week Follow-Up
Population: Analysis only includes those participants who responded to the measure at 1-Week Follow-Up (DA=27, no-DA=28, Total=55).
Measure: Mean (Standard Deviation); unit: years
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 27 | 28
years | 10.17 (7.14) | 9.7 (9.8)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Satisfaction With Life
Description: Satisfaction with Life Scale, intended to measure respondents' perceived global life satisfaction. Out of 0-30 scale. Higher scores indicate higher satisfaction with life.
Time Frame: 1-Month Follow-Up
Population: Analysis only included those participants who completed the measure at 1-Month Follow-Up (DA=26, no=DA=30, Total=56).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 30
units on a scale | 27.9 (5.7) | 22.9 (6.9)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Quality of Life -- Health Rating
Description: Responses to the question: "On a scale of 0 to 100 (0 is the worst health imaginable, 100 is the best health imaginable) what would you rate your health today?"
Time Frame: Baseline
Population: Analysis included only those participants who completed the measure at baseline (DA=46, no-DA=50, Total=96).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 46 | 50
units on a scale | 55.8 (24.0) | 43.1 (24.5)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Quality of Life -- Health Rating
Description: as for outcome 23
Time Frame: 1-Month Follow-Up
Population: Analysis included only those participants who completed measure at 1-Month (DA=26, no-DA=30, Total=56).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 30
units on a scale | 81.0 (3.7) | 69.1 (3.5)
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Preferred Treatment: Number of Patients Predicting They Will Choose LVAD
Description: Number of patients forecasting that they will choose LVAD treatment (before their actual decision), measured using a binary score representing yes (1) or no (0) indicating whether a patient predicted they would choose LVAD as a preferred treatment for their advanced heart failure.
Time Frame: Baseline
Population: Analysis only includes participants who responded to the question at baseline (DA=46, no-DA=50, Total=96).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 46 | 50
Participants | 28 | 31

26. Secondary Outcome: Number of Patients Whose Preferred Treatment Was LVAD
Description: Number of patients who definitively choose LVAD treatment, measured using a binary score representing yes (1) or no (0) indicating whether the patient chose LVAD as a preferred treatment for their advanced heart failure.
Time Frame: 1-Week Follow-Up
Population: Analysis only includes participants who responded to the question at 1-Week (DA=28, no-DA=33, Total=61).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 28 | 33
Participants | 21 | 26
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Number of Patients Whose Preferred Treatment Was LVAD
Description: as for outcome 26
Time Frame: 1-Month Follow-Up
Population: Analysis only includes participants who responded to the question at 1-Month (DA=26, no-DA=32, Total=58).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 32
Participants | 22 | 25
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Number and Percentage of Patients Who Filled Out an Advanced Directive
Description: Number and percentage of patients who filled out an Advanced Directive, using a binary measure indicating whether a respondent has filled out an advanced directive (1) or not (0).
Time Frame: 1-Month Follow-Up
Population: Analysis only includes participants who responded to the question (DA=25, no-DA=27, Total=52).
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 25 | 27
Participants | 17 | 12
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.12, Fisher Exact

29. Secondary Outcome: Usability and Acceptability: Helped me Understand my Options for Dealing With Heart Failure.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 35 | 0
Participants
  Strongly Agree | 19 | 0
  Agree | 11 | 0
  Neutral | 4 | 0
  Disagree | 1 | 0
  Strongly Disagree | 0 | 0

30. Secondary Outcome: Usability and Acceptability: Learned Something New That I Didn't Know Before.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 35 | 0
Participants
  Strongly Agree | 20 | 0
  Agree | 9 | 0
  Neutral | 5 | 0
  Disagree | 1 | 0
  Strongly Disagree | 0 | 0

31. Secondary Outcome: Usability and Acceptability: Would Recommend to Others.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: Analysis included only those participants who completed this question in the 1-Day Follow-up measure, which was 37 patients in the DA group. The no-DA group did not receive the measure.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 37 | 0
Participants
  Yes | 34 | 0
  Unsure | 3 | 0
  No | 0 | 0

32. Secondary Outcome: Usability and Acceptability: Held my Interest.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 37 | 0
Participants
  Yes | 34 | 0
  Unsure | 2 | 0
  No | 1 | 0

33. Secondary Outcome: Usability and Acceptability: Helps Someone Make an Informed Decision.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 35 | 0
Participants
  Yes | 33 | 0
  Unsure | 2 | 0
  No | 0 | 0

34. Secondary Outcome: Usability and Acceptability: Helped me to Think About Aspects of Heart Failure Treatment That Matter Most to me.
Description: Measures the usability and acceptability of the decision aid 1 day after receiving the decision aid tool
Time Frame: 1 Day Follow-up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 35 | 0
Participants
  Yes | 30 | 0
  Unsure | 4 | 0
  No | 1 | 0

35. Secondary Outcome: Participants' Control Preferences Over Treatment Decision-Making
Description: This data is based on responses to a 1-item questionnaire (i.e. not a scale). Scores are calculated by counting the frequency of matches in patient-reported preferences at two time points.
Time Frame: Baseline
Population: Analysis only included participants who completed the measure at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 46 | 49
Participants
  Patient made final decision | 5 | 5
  Patient, after seriously considering doctor opinio | 15 | 17
  Doctor and patient shared responsibility | 18 | 21
  Doctor made decision after considering patient opi | 5 | 4
  All decisions left to doctor | 3 | 2
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.98, Fisher Exact

36. Secondary Outcome: Participants' Control Preferences Over Treatment Decision-Making
Description: This data is based on responses to a 1-item questionnaire (i.e. not a scale). Scores are calculated by counting the frequency of matches in patient-reported preferences at two time points (baseline and 1-month follow-up).
Time Frame: 1-Month
Population: Analysis only included participants who completed the measure at baseline, minus participants lost to attrition between baseline and 1-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Number analyzed (Participants) | 26 | 30
Participants
  Patient made final decision | 3 | 1
  Patient, after seriously considering doctor opinio | 10 | 18
  Doctor and patient shared responsibility | 10 | 8
  Doctor made decision after considering patient opi | 1 | 3
  All decisions left to doctor | 2 | 0
Statistical Analysis 1: Comparison: LVAD Decision Aid vs No LVAD Decision Aid; Test type: Superiority; p = 0.20, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events data were monitored and assessed over a period of 3 years, from the beginning of Aim 1 to the end of Aim 2 of the study, using patient data files kept by LVAD coordinators at participating clinics and given to us securely.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, did not differ from the clinicaltrials.gov definitions.
Arm/Group | LVAD Decision Aid | No LVAD Decision Aid
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51
Other Adverse Events (participants affected / at risk) | 0/47 | 0/51

LIMITATIONS AND CAVEATS:
No significant limitations to report. One consideration is that because we tested for efficacy at sites with established LVAD programs, results may not be generalizable to other less well-run programs, where effect sizes may be even greater.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes